CLINICAL TRIAL: NCT00130338
Title: An Open-label Extension to Evaluate the Efficacy and Safety of Rivastigmine Capsules in Patients With Probable Vascular Dementia
Brief Title: Rivastigmine Capsules in Patients With Probable Vascular Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713BIA05E1
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Vascular Dementia
Keywords: Dementia; Vascular; Rivastigmine; Stroke; Memory loss
MeSH Terms: conditions — Dementia, Vascular; Dementia; Stroke; Memory Disorders | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine

SUMMARY:
The goal of this research study is to evaluate, in the open-label extension phase, the effectiveness, tolerability and safety of rivastigmine capsules in males and females between the ages of 50 and 85 years old with probable vascular dementia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who complete the double-blind treatment phase or those who have dropped out early in the study, but have returned for all the remaining scheduled efficacy assessments (retrieved drop-out patients) without significant protocol violations are eligible to participate.

Exclusion Criteria:

* Retrieved drop-out patients, who have been treated with other cholinergic drugs during the past 4 weeks

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2002-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of rivastigmine for up to 52 weeks of treatment in patients with VaD and probable VaD

SECONDARY OUTCOMES:
52 week's treatment with rivastigmine on cognition, activities of daily living, behavior and clinical staging in patients with VaD and probable VaD